CLINICAL TRIAL: NCT03889002
Title: Health Indicators, Functioning and Health Care Services in Youths and Adults With Intellectual Disabilities. A Cross-sectional Multicentre Study.
Brief Title: North Health in Intellectual Disability
Acronym: NOHID
Status: Completed | Type: Observational
Sponsor: University Hospital of North Norway (Other)
Collaborators: Norwegian Extra Foundation for Health and Rehabilitation (Other); The Norwegian Association for Persons with Developmental Disabilities (Unknown); University of Tromso (Other); Norwegian University of Science and Technology (Other); Research Centre for Habilitation and Rehabilitation Models and Services (Unknown); Norwegian Centre for Ageing and Health (Other)
Responsible Party: Sponsor
Other Study IDs: 2017/811
Record Dates: First submitted 2019-03-04; First posted 2019-03-25 (Actual); Last update posted 2020-04-06 (Actual); Status verified 2019-03

CONDITIONS: Intellectual Disabilities (F70-F79)
Keywords: Intellectual disabilities; Health indicators; Functioning; Health care services
MeSH Terms: conditions — Intellectual Disability

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Intellectual disability (ID) is a diagnosis characterized by significant limitations both in intellectual functioning and in adaptive behavior as expressed in conceptual, social and practical adaptive skills. The disability originates before age 18 years. People with IDs will often require health- and social services throughout their lifetimes. Studies report worse health among people with IDs compared to the general population, in addition to more unmet healthcare needs and more difficulty accessing healthcare. There are also concerns about low levels of physical activity in this population.

In general health surveys in Norway do not include people with intellectual disabilities, and studies of health indicators in this group are largely lacking. Further, the unique organization of services for this group in Norway calls for specific research efforts. This project will use multinational health indicators for youths and adults with IDs in a biopsychosocial context in attempt to identify unmet health care needs to improve services. In addition to a description of the health indicators, the objective of this project is delimited to assess the health determinant physical activity level in association with body mass index (BMI) and functioning.

DETAILED DESCRIPTION:
People with IDs are experiencing more illnesses and approximately 80% of adults 50 years or older have multimorbidities. To improve services, information about health care provision should be complemented with knowledge about the health situation and functioning in a community-based setting.

The main objectives of this study are to describe health indicators in a Norwegian population of youths and adults with IDs in relation to age, and to assess the associations between the health determinant physical activity and body mass index, physical function, activities and social participation in youths and adults with IDs.

Assessments of physical and mental health indicators, and aspects of activities and social participation according to International Classification of Functioning, Disability and Health (ICF), in relation to health determinants and unmet healthcare needs in a cross-sectional health screening survey.

The prevalence of suitable health indicators will be compared to studies in this area and from the following Norwegians population based studies: the "Tromsø-study", the "HUNT" study and the "NORSE study".

The following articles will be published as part of this project:

1. A feasibility study of the use of tests like the Short Physical Performance Battery.
2. An overview of the health indicators among youths and adults with intellectual disabilities in Norway, in relation to age groups.
3. Presentation of levels and predictors for physical activity, as well as body mass index, in youths and adults with IDs.
4. Presentation of functioning (daily activities and work) in association to levels of physical activity.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of intellectual disability
* Age 16 or older and providing consent to participate.

Exclusion Criteria:

-

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Persons with intellectual disabilities and registered services in the municipalities in two regions localised in the north and middle of Norway will be invited to participate in the study.
Sampling Method: Probability Sample
Enrollment: 214 (Actual)
Dates: Start 2017-10-01 (Actual); Primary Completion 2019-12-09 (Actual); Study Completion 2019-12-09 (Actual)

PRIMARY OUTCOMES:
Health indicators in a Norwegian population of youths and adults with intellectual disabilities. | Baseline
  Health indicators as measured by The POMONA Checklist of Health Indicators (P15). The health indicators include measures of socio-demographics, Health status, Health determinants and Health systems.Physical Activity is defined as a Health determinant in this study in accordance With the POMONA Health indicator classification.

SECONDARY OUTCOMES:
Communication Function Classification System (CFCS). | Baseline
  The CFCS is a 5-category rating system. Where Level 1 is best and Level 5 worst.
The Community Integration Questionnaire (CIQ). | Baseline
  The scale contains 15 items to assess social role limitations and community interactions in persons With Health disorders. The items are scored on a likert-type scale. The total scale range fraom 0-29 where 29 is Maximum community integration.
The Coherence of social care scale. | Baseline
  The Coherence of social care scale measures the coherence of social care and the stability of services in general. The scale uses a responscale from 1-4 (higher is better)
The Short Physical Performance Battery (SPPB). | Baseline
  The SPPB measures physical functioning like balance, gait and muscular functioning. Total scale range from 0-12 (higher score indicate better functionin).
The Timed Up and GO (TUG). | Baseline
  The TUG measures Balance, gait and general functioning. The time one person use to get up from a Chair, walk 3 meters and then return back to the Chair is measured in Seconds. Less time is better functioning.
One-legged Stance test | Baseline
  The One-legged Stance test measures balance. The time in Seconds of how long a person can Balance on one legg is measured. Longer time is better functioning.
The Gross Motor Function Classification Scale (GMFCS). | Baseline
  The GMFCS measures motor functioning. It is a 5-category rating scale where 1 is most able and 5 is most Limited functioning.
Body mass index (BMI) | Baseline
  BMI is calculated by measuring height and weight.
Overarm circumference. | Baseline
  Overarm circumference is measured.
Measuring Bloodpressure. | Baseline
  Systolic and diastolic bloodpressure are measured.
Waist circumference | Baseline
  Waist circumference is measured.

CONTACTS AND LOCATIONS:
Overall Officials: Audny Anke, MD, professor, Principal Investigator — University Hospital of North Norway, Sykehusveien 38, 9038 Tromsø
Locations (1):
- University Hospital of North Norway, Tromsø, Norway

REFERENCES:
- [Derived] Olsen MI, Sondenaa E, Langballe EM, Halvorsen MB, Wilhelmsen P, Bautz-Holter E, Anke A. Use of health and dental care services in adults with intellectual disability in relation to age and intellectual disability levels. J Intellect Dev Disabil. 2023 Jun;48(2):172-183. doi: 10.3109/13668250.2022.2109823. Epub 2022 Oct 18. PMID 39815906